CLINICAL TRIAL: NCT05375708
Title: A Multicenter Phase II Randomized Trial to Evaluate Systemic Therapy Versus Systemic Therapy in Combination with Stereotactic Radiotherapy in Patients with Metastatic Colorectal Cancer
Brief Title: Systemic Therapy in Combination with Stereotactic Radiotherapy in Patients with Metastatic Colorectal Cancer Up to 10 Metastatic Sites
Acronym: SIRIUS
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Pilot study findings pointed to a overhaul in study design
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Guus Bol, Principal investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL76444.041.21
Record Dates: First submitted 2022-04-05; First posted 2022-05-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer; Oligometastatic Disease
Keywords: Metastatic colorectal cancer; Image guided radiation; MR guided therapy; Oligometastatic / polymetastatic cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; Maintenance; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systemic maintenance therapy (Active Comparator)
  Interventions: Drug: Maintenance therapy (CAP-B or 5-FU/LV plus bevacizumab.)
- Systemic maintenance therapy in combination with stereotactic body radiation therapy (SBRT) (Experimental)
  Interventions: Radiation: Stereotactic body radiation therapy (SBRT); Drug: Maintenance therapy (CAP-B or 5-FU/LV plus bevacizumab.)

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy (SBRT) — Patients will receive a single fraction of 15 Gy to each of the macroscopic tumor sites including the primary tumor if still in situ. All lesions are treated. The treatment will be delivered in an image-guided way, either on a conventional linear accelerator (LINAC) or a MR-LINAC, whichever has the best targeting according to the treating radiation oncologist.
  Arms: Systemic maintenance therapy in combination with stereotactic body radiation therapy (SBRT)
Drug: Maintenance therapy (CAP-B or 5-FU/LV plus bevacizumab.) — CAP + bevacizumab (following CAPOX-B) Bevacizumab 7.5mg/kg i.v. on day 1 and 1250 mg/m2 of capecitabine, orally twice daily on days 1-14 if age is <70 years and 1000 mg/m2 of capecitabine, orally twice daily on days 1-14 if age is higher than 70 years. CAP + bevacizumab is repeated every three weeks.
  5-FU/LV + bevacizumab (following FOLFOX-B) Bevacizumab 5.0mg/kg i.v. together with leucovorin 400 mg/m2 i.v. bolus 5FU 400 mg/m2 all on day 1. Followed by continuous infusion of 5-fluorouracil 2400 mg/m2 in 46 hours. 5-FU + bevacizumab is repeated every two weeks.
  5-FU/LV + bevacizumab (following FOLFOXIRI-B) Bevacizumab 5.0mg/kg i.v. together with leucovorin 400 mg/m2 i.v. all on day 1. Followed by continuous infusion of 5-fluorouracil 3200 mg/m2 in 46 hours. 5-FU + bevacizumab is repeated every two weeks.
  When S1 is used a replacement for fluoropyrimidine therapy it is administered in a dose of 30mg/m2 twice daily on days 1-14. S1 is repeated every three weeks.

SUMMARY:
A small number of colorectal cancer patients with limited oligometastases may be candidates for local treatment of metastases (e.g., resection, ablation). However, it is unclear if patients with more extensive metastatic disease benefit from local therapies to control visible metastasis.

The purpose of this study is to assess the impact of stereotactic body radiation therapy (SBRT) in combination with systemic therapy compared to systemic therapy alone on safety and efficacy in patients with metastatic colorectal cancer (mCRC) and ≤10 metastases.

DETAILED DESCRIPTION:
The addition of stereotactic body radiation therapy (SBRT) to metastases in a limited unresectable metastatic setting might improve progression-free survival (PFS). The success of the addition of local treatments in mCRC patients depends largely on: control of microscopic disease, diagnostic accuracy of macroscopic disease and effective treatment of all detected metastases with limited additional toxicity to surrounding tissues. Until shortly, the use of SBRT was possible to a limited number of locations due to target movement or toxicity to surrounding radiosensitive structures. With the introduction of MRI-guided radiotherapy these limitations have been largely reduced due to the possibility to make a daily new treatment plan based on MRI-visualized anatomy. This allows the use of smaller margins for uncertainty with less healthy tissues in the radiation field. Thereby, a broader application of SBRT to add local control to metastases became possible.

This study is an open-label, multicenter, randomized phase II screening trial assessing the impact of SBRT in combination with systemic therapy compared to systemic therapy alone on safety and efficacy in patients with mCRC and ≤10 metastases with no option of local treatment with curative intent and with stable disease or partial response after treatment of CAPOX-B, FOLFOX-B or FOLFOXIRI-B.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the prospective Dutch colorectal cancer cohort (PLCRC)
* Intention at start of palliative systemic therapy to receive six maximum tolerated dose (MTD) cycles of CAPOX-B or eight MTD cycles of FOLFOX-B or FOLFOXIRI-B.
* Ten or less metastases as determined by the university medical center Utrecht (UMCU) central review
* Stable disease or partial response after initial chemotherapy according to RECIST 1.1 criteria.
* Expected adequacy of follow-up
* World Health organization (WHO) performance status 0-1
* Life expectancy >12 weeks
* Adequate organ functions at start of initial therapy, as determined by normal bone marrow function (Hb≥6.0 mmol/L, absolute neutrophil count ≥1.5 x 10^9/L, platelets ≥100 x 10^9/L), renal function (serum creatinine ≤ 1.5x upper limit of normal (ULN) and creatinine clearance, Cockcroft formula, ≥30 ml/min) and liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases)
* Written informed consent (SIRIUS)

Exclusion Criteria:

* Less than three cycles of CAPOX-B or four cycles of FOLFOX-B or FOLFOXIRI-B (dose reductions allowed).
* More than six cycles of CAPOX-B or eight cycles of FOLFOX-B of FOLFOXIRI-B.
* Possible treatment with curative intent according to local tumor board
* Substantial overlap with a previously treated radiation volume. Previous radiotherapy is allowed as long as the composite plan meets dose constraints herein.
* Not amenable for radiotherapy (e.g. peritonitis carcinomatosa)
* Previous systemic treatment for metastatic disease; prior adjuvant treatment for stage II/III colorectal cancer when given >6 months before the start of initial systemic treatment is allowed.
* Serious comorbidity or any other condition preventing the safe administration of treatment (including both systemic treatment and radiation)
* Pregnant or lactating women
* Other malignancy interfering with prognosis
* Any concomitant experimental treatment.
* Contra-indication MR-LINAC (pacemaker or implantable cardioverter-defibrillator)
* Microsatellite instability or deficient mismatch repair tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2031-06-01 (Estimated); Study Completion 2034-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, an average of 24 months
  Defined as time from randomization to progression of disease or death, whichever occurs first. Progression of disease is based on tumor response as observed on radiographic imaging according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Accrual rate as assessed by the number of patients included in the study compared to the expected accrual rate. | Through study completion, an average of 24 months
  We expect to include 93 patients in 24 months. The expected accrual rate in this study is, therefore, around 4 patients per month. Information for the accrual rate is used from the total accrual rate, the accrual rate in each study center and screening failures.
Treatment success rate | Through study completion, an average of 24 months
  Dose intensity of SBRT based on the number of patients that receive more than 90% of the planned dose on all lesions in 95% of the planned target volume (PTV).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, an average of 24 months
  This will be based on the number of patients with SBRT related toxicity, defined as newly developed grade 2 toxicity of specific interest and grade 3-4 toxicity since randomization according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Overall survival | Up to 72 months
  Defined as time from randomization to death of any cause.
Comparing changes on health-related quality of life based on summary score of Quality of Life Questionnaire-Core30 (QLQ-C30) from baseline and 3-monthly timepoints. | Through study completion, an average of 24 months
  EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score is better level of functioning.
Comparing changes on health-related quality of life based on summary score of Quality of Life Questionnaire-Core29 (QLQ-C29) from baseline and 3-monthly timepoints. | Through study completion, an average of 24 months
  EORTC QLQ-C30 is a 29-item questionnaire to assess the overall quality of life in cancer patients. All questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score is better level of functioning.
Comparing changes from health-related quality of life based on summary score of Multidimensional Fatigue Inventory (MFI-20) from baseline and 3-monthly timepoints. | Through study completion, an average of 24 months
  MFI is a validated 20-item, self-reported instrument designed to measure fatigue in the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The respondent is asked to mark an 'X' in 1 of 5 boxes arranged linearly where 1 is 'Yes, that is true' and 5 is 'No, that is not true.' Each subscale consists of 4 items, 2 indicative for fatigue and 2 contraindicative. For the indicative questions, a high score indicates a high fatigue level and low scores indicate a low fatigue levels. Conversely, for the contraindicative questions a high score indicates a low fatigue level and a low score indicates a high fatigue level. Overall, respondents are rated on a scale of 0 (no fatigue) to 7 (high fatigue).
Pattern of reccurence according to RECIST 1.1: New metastatic lesions, progression of existing lesions or a combination. | Through study completion, an average of 24 months
  New metastatic lesions, progression of existing lesions or a combination of both new metastatic lesions and progression of existing lesions based on radiographic imaging according to RECIST 1.1
Time to treatment failure | Through study completion, an average of 24 months
  Defined as the time of randomization to failure of treatment. If radiologically visible metastatic lesions before systemic therapy are no longer visible at randomization (vanishing lesions) and recurrence of vanishing lesions occurs in patients in the experimental arm without progression of other lesions, this is not yet determined as failure of treatment; additional local therapy is highly encouraged on these lesions (to the discretion of the local investigator). When progression of existing lesions or new lesions occur, it will be determined as failure of treatment.
Tumor response | Through study completion, an average of 24 months
  Based on radiographic imaging according to the RECIST 1.1 criteria.
Depth of response | Through study completion, an average of 24 months
  Based on radiographic imaging

CONTACTS AND LOCATIONS:
Overall Officials: Guus Bol, Dr., Principal Investigator — UMC Utrecht; Martijn Intven, Dr., Principal Investigator — UMC Utrecht; Miriam Koopman, Prof. Dr., Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Meander Medical Centre, Amersfoort, Utrecht
  - St. Antonius, Utrecht, Utrecht
  - Diakonessenhuis, Utrecht, Utrecht
  - UMC Utrecht, Utrecht, Utrecht